CLINICAL TRIAL: NCT03463889
Title: Gallium-68 Prostate Specific Membrane Antigen (68Ga-PSMA) PET for Imaging of Thyroid Cancer: A Feasibility Study
Brief Title: Gallium-68 Prostate Specific Membrane Antigen PET in Diagnosing Patients With Thyroid Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Robert Flavell, MD, PhD, Asst Professor in Residence, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 172016; NCI-2018-00055 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-02-09; First posted 2018-03-13 (Actual); Results first posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Thyroid Gland Carcinoma
MeSH Terms: conditions — Thyroid Neoplasms | interventions — gallium 68 PSMA-11; Magnetic Resonance Spectroscopy; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (Gallium Ga 68-labeled PSMA-11, PET/MRI) (Experimental): Participants receive 68Ga-PSMA IV over 1-2 minutes and then undergo PET/MRI 60 minutes after injection. Patients may undergo a second PET/MRI 2-6 months after completion of first scan.
  Interventions: Drug: Gallium Ga 68-labeled PSMA-11; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography (PET)

INTERVENTIONS:
Drug: Gallium Ga 68-labeled PSMA-11 — Given IV
  Other Names: 68Ga-HBED-CC-PSMA; 68Ga-PSMA-11; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; Ga-68 labeled PSMA-11; Gallium Ga 68 PSMA-11
Procedure: Magnetic Resonance Imaging — Undergo MRI in combination with PET
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI; MRI Scan; Nuclear Magnetic Resonance Imaging (NMRI); Nuclear Magnetic Resonance (NMR) Imaging; NMRI
Procedure: Positron Emission Tomography (PET) — Undergo PET in combination with MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This pilot clinical trial studies how well Gallium-68 prostate specific membrane antigen positron emission tomography (PET) work in diagnosing patients with thyroid cancer. Diagnostic procedures, such as 68Ga-PSMA PET, may more accurately diagnose thyroid cancer and find out how far the disease has spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility and utility of Gallium Ga 68-labeled PSMA-11 (68Ga-PSMA) PET imaging in patients with thyroid cancer.

SECONDARY OBJECTIVES:

I. To assess the correlation between targeted molecular uptake of 68Ga-PSMA PET in thyroid cancer compared to areas identified as tumor by radioiodine uptake (in well-differentiated cancers) or fludeoxyglucose F-18 (18F-FDG) uptake (in poorly differentiated and/or radioiodine-negative cancers).

II. To determine and compare the sensitivity and specificity of 68Ga-PSMA PET to (18F-FDG) PET and/or radioiodine scintigraphy.

TERTIARY OBJECTIVES:

I. To determine if 68Ga-PSMA PET uptake is related to tumor differentiation and PSMA staining in tissue pathology when available.

II. To determine the correlation between standardized uptake value maximum (SUVmax) of target thyroid cancer lesions on 68Ga-PSMA PET and serum thyroglobulin levels.

OUTLINE:

Participants receive 68Ga-PSMA intravenously (IV) over 1-2 minutes and then undergo PET/MRI 60 minutes after injection. Patients may undergo a second PET/MRI 2-6 months after completion of first scan.

ELIGIBILITY:
Inclusion Criteria:

* History of thyroid cancer
* Whole body 18F-FDG PET/computed tomography (CT) or I-131 scintigraphy within the past 90 days of the scheduled 68Ga-PSMA PET demonstrating uptake
* Creatinine =< 3.0 mg/dL
* Ability to understand a written informed consent document, and the willingness to sign it

Exclusion Criteria:

* Patients who have had active infection within 15 days of study enrollment that may be considered to interfere with 68Ga-PSMA PET imaging by the study investigators
* Patients who are unable to have placement of intravenous line access
* Pregnant or breastfeeding women
* Patients not capable of undergoing a PET/MRI study due to weight, claustrophobia, or inability to lie still for the duration of the exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Flavell, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic (Gallium Ga 68-labeled PSMA-11, PET/MRI)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (Gallium Ga 68-labeled PSMA-11, PET/MRI)
Number analyzed (Participants) | 12
Age, Customized [Count of Participants; unit: Participants]
  40-49 years old | 2
  50-59 years old | 2
  60-69 years old | 4
  70-79 years old | 3
  80-89 years old | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 12
Years from initial diagnosis to study imaging [Median (Full Range); unit: years] | 3 [0 to 28]

OUTCOME MEASURES:

1. Primary Outcome: Number of 68Ga PSMA-11 PET-positive Lesions
Description: The number of 68Ga PSMA-11 PET-positive lesions detected by staging scans will be descriptively reported.
Time Frame: Up to 24 months
Population: One patient with qualifying FDG PET/CT underwent surgical procedures prior to undergoing [68Ga]Ga-PSMA-11 PET/MRI and was therefore excluded from the analysis due to lack of comparability
Measure: Number; unit: lesions
Arm/Group | Diagnostic (Gallium Ga 68-labeled PSMA-11, PET/MRI)
Number analyzed (Participants) | 11
lesions | 28

2. Primary Outcome: Number of Overall Detected Thyroid Cancer Lesions
Description: The number of overall thyroid cancer lesions detected by standard staging scans will be descriptively reported
Time Frame: Up to 24 months
Population: as for outcome 1
Measure: Number; unit: lesions
Arm/Group | Diagnostic (Gallium Ga 68-labeled PSMA-11, PET/MRI)
Number analyzed (Participants) | 11
lesions | 43

3. Primary Outcome: Mean Standardized Uptake Value Maximum of Gallium-68 PSMA (SUVmax)
Description: The mean and standard deviation for SUVmax across all lesions across all patients will be reported.
Time Frame: Up to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Diagnostic (Gallium Ga 68-labeled PSMA-11, PET/MRI)
Number analyzed (Participants) | 11
Ratio | 8.5 (5.7)

4. Secondary Outcome: Sensitivity of Gallium-68 PSMA for the Detection of Thyroid Cancers
Description: For each lesion detected on 18F-FDG PET or radioiodine scintigraphy (131I), the presence or absence of 68Ga-PSMA-11 uptake will be reviewed and tabulated. Presence on either 131I and 18F-FDG will be considered true positive disease. If additional lesions are detected on 68Ga-PSMA-11 as compared to 18F-FDG or 131I, the lesions will be characterized as either true or false positives in comparison to the appearance of the lesion on conventional imaging (thyroid ultrasound, CT and MRI). The gold standard for an individual lesion will be FDG or 131I, if the individual lesion is positive on either imaging study. If the lesions are not seen on either FDG or 131I, then consensus reading of conventional imaging will be performed to determine true and false positives lesions. Point estimate of the true positive rate will be calculated.
Time Frame: Up to 24 months
Population: as for outcome 1
Measure: Number; unit: proportion of participants
Arm/Group | Diagnostic (Gallium Ga 68-labeled PSMA-11, PET/MRI)
Number analyzed (Participants) | 11
proportion of participants | .65

5. Secondary Outcome: Specificity of Gallium-68 PSMA for the Detection of Thyroid Cancers
Description: Specificity is the agents ability to exclude the disease when the disease is absent. For each lesion detected on 18F-FDG PET or radioiodine scintigraphy (131I), the presence or absence of 68Ga-PSMA-11 uptake will be reviewed and tabulated. Presence on either 131I and 18F-FDG will be considered true positive disease. If additional lesions are detected on 68Ga-PSMA-11 as compared to 18F-FDG or 131I, the lesions will be characterized as either true or false positives in comparison to the appearance of the lesion on conventional imaging (thyroid ultrasound, CT and MRI). The gold standard for an individual lesion will be FDG or 131I, if the individual lesion is positive on either imaging study. If the lesions are not seen on either FDG or 131I, then consensus reading of conventional imaging will be performed to determine true and false positives lesions. Point estimate of the true negative rate will be reported.
Time Frame: Up to 24 months
Population: as for outcome 1
Measure: Number; unit: proportion of participants
Arm/Group | Diagnostic (Gallium Ga 68-labeled PSMA-11, PET/MRI)
Number analyzed (Participants) | 11
proportion of participants | 1.00

ADVERSE EVENTS:
Time Frame: Up to 6 months
Description: Only grade 3 and higher adverse events were recorded
Arm/Group | Diagnostic (Gallium Ga 68-labeled PSMA-11, PET/MRI)
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
Study closed earlier than expected due to lack of funding. Due to the small sample size, comparative sub-group analyses could not be performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT03463889/Prot_SAP_000.pdf